CLINICAL TRIAL: NCT01629056
Title: The Contact-PVI Study - Does Assessment of Tissue Contact During RF Ablation Using the St. Jude Medical™ Ensite™ Contact™ System Increase Rates of Long-term Pulmonary Vein Isolation? A Prospective Randomised Study
Brief Title: The Contact PVI Study: Use of Tissue Contact Data to Guide Atrial Fibrillation Ablation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 77431/244334/1/228; 11/SC/0398 (Other: Oxford C NRES Committee South Central)
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; ablation; contact
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contact ECI active (Active Comparator): Contact ECI active
  Interventions: Procedure: ablation
- Contact information deactivated (Placebo Comparator): RF ablation without contact data
  Interventions: Procedure: RF ablation

INTERVENTIONS:
Procedure: ablation — RF ablation to the left atrium of the heart, guided by ECI-contact information (active arm)
  Other Names: Irrigated RF ablation; RF ablation; Percutaneous transvenous catheter ablation
  Arms: Contact ECI active
Procedure: RF ablation — RF ablation to the left atrium of the heart, without the use of ECI-contact information (control arm)
  Other Names: Irrigated RF ablation; Percutaneous transvenous catheter ablation
  Arms: Contact information deactivated

SUMMARY:
This study aims to investigate the benefit of a new impedance-based computer software application during routine catheter ablation for atrial fibrillation, to see if this information improves short and long term electrical disconnection of the pulmonary veins. This study will be a single blind prospective randomised control trial in patients undergoing AF ablation. Study participants will be randomly assigned to undergo parts of their pulmonary vein ablation with, and parts of their ablation without tissue contact data displayed for the doctor performing the ablation to see. The pulmonary veins will then be studied at the end of the procedure, and at any repeat procedure in the future, to look for a difference in the recovery rate of the ablations performed using contact data, compared to those ablations performed without the use of this contact data. If a reduction in tissue recovery is achieved through the use of this tissue contact data, it may lead in the future to a reduced need for repeat ablation procedures, and better outcomes for patients.

The investigators hypothesise that the use of the Ensite™ Contact™ ECI data will reduce the recovery of conduction, and promote long-term pulmonary vein isolation in patients undergoing left atrial ablation for atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is undergoing de novo pulmonary vein isolation procedure.
2. Participant is willing and able to give informed consent for participation in the study.
3. Male or Female, ≥18 years of age.

Exclusion Criteria:

1. Previous percutaneous or open surgical procedure involving the left atrium
2. Pregnancy (current or currently planning)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-02-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the proportion (%) of pulmonary vein pairs found to be reconnected electrically to the left atrium at a subsequent redo ablation procedure | 6 months

SECONDARY OUTCOMES:
Proportion of acute venous electrical reconnections | acute (intra-procedure)
  proportion of pulmonary veins found to be electrically reconnected to the left atrium at the end of the index procedure
touch-up ablation requirements | acute (intra-procedure)
  proportion of veins requiring additional ablation after initial successful isolation, at the end of the index procedure
procedure time | acute
  duration of procedure
RF time | acute (intra-procedure)
  total amount of radiofrequency ablation required
anatomical location of reconnections at repeat procedure | at repeat ablation procerdure (6-12 months post index ablation procedure)
  anatomical location of electrical reconnections in pulmonary vein antra, as measured at a repeat ablation procedure
amount of RF required to achieve re-isolation at repeat ablation procedure | at repeat ablation procedure (6-12 months post-index ablation procedure)
  total time of RF delivery required to re-isolate the reconnected pulmonary veins at a repeat ablation procedure
complications | acute and subacute (intra-procedure, and during entire follow-up period)
  procedure-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Jones, MBBS, Principal Investigator — Oxford University Hospitals NHS Trust; Tim R Betts, MbCHb PhD, Study Director — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Headington, Oxfordshire, United Kingdom